CLINICAL TRIAL: NCT02863978
Title: Preliminary Study to the Conception of a Non-invasive Neonatal Monitoring System With Development of a Database
Acronym: Digi-NewB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rennes University Hospital (Other)
Collaborators: European Union (Other); GCS Hôpitaux Universitaires Grand-Ouest (Unknown); Rennes 1 University (Unknown); Tampere University of Technology (Other); Voxygen Health (Unknown); INESC TEC Porto (Unknown); National University of Ireland, Galway, Ireland (Other); Synchrophi Systems Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 35RC16_9714; 2016-A00993-48 (Other: ID-RCB)
Record Dates: First submitted 2016-08-03; First posted 2016-08-11 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Infant, Premature
Keywords: Sepsis; Neonates; Cardio-respiratory maturation; Neurobehavioral maturation
MeSH Terms: conditions — Premature Birth; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Digi-NewB Cohort (Experimental): Multimodal signal acquisitions
  Interventions: Other: Multimodal signal acquisitions

INTERVENTIONS:
Other: Multimodal signal acquisitions — Cardiac and respiratory signals are collected from the clinical monitoring routinely gathered in hospital neonatal units.
  Movement quantification and baby's sounds are extracted thanks to a dedicated system which will collect images and sound with microphones and cameras.

SUMMARY:
Each year, 300 000 new borns are hospitalised in neonatology units in Europe. This period is very sensitive as newborns are exposed to a high risk of morbidity and mortality, with severe impact on neuro-developmental prognostic. The Rennes University Hospital was granted a specific funding from the European Union in the framework of the Horizon 2020 programme (Call PERSONALISING HEALTH AND CARE 2015-single-stage - Grant Agreement Number 689260) to develop the Digi-NewB project. This project aims to develop innovative non-invasive monitoring tools to support decision making in health. Such tools include a new generation of real time monitoring in neonatology using composite indices made of cardio-respiratory variables, movements, sounds, and clinical data. The Digi-NewB cohort aims to gather all physiological data relevant for the creation of the composite indices.

DETAILED DESCRIPTION:
The database will be used to answer the following specific objectives, with priority given to the two first ones (sepsis and maturation) :

1. Early diagnosis of sepsis for the following cases : Late onset sepsis of premature newborns, materno-fœtal sepsis, and newborn infection by chorioamnionitis
2. Cardio-respiratory and neurobehavioral maturation (movements, sleeping cycles)
3. Influence of environmental factors and developmental care on selected parameters
4. Influence on care organisation of the possibility to access videos and movement analyses by medical teams
5. Influence of glycemia on selected parameters
6. Influence of neurological lesions and broncho-pulmonary dysplasia on selected parameters
7. Indices correlation with medical images MRI (T1, T2, diffusion, Arterial Spin Labelling) from neonatal units and with health evaluated after 1 and 2 years with the Ages & Stages Questionnaires (ASQ)
8. Evaluation of the acquisition system's user-friendliness

ELIGIBILITY:
Inclusion Criteria:

* Newborn hospitalised in the neonatology services of participating hospitals
* One of the legal representatives gave its signed agreement to take part to the study
* New born aged of less than 6 weeks in corrected term

Exclusion Criteria:

* No signed agreement from the legal representative

Max Age: 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 746 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
Number of newborns in neonatology unit | Four years

SECONDARY OUTCOMES:
Infection/Sepsis | During the stay in neonatal unit, up to 10 weeks
  Identification of late onset sepsis of premature newborns, materno-fœtal sepsis, and newborn infection by chorioamnionitis
Maturation | During the stay in neonatal unit, up to 10 weeks
  Quantification of maturation, i.e. evaluation of cardio respiratory rates and neurobehavioral maturation
Influence of environment and developmental care | During the stay in neonatal unit, up to 10 weeks
  Measure of impact of access to new variables (maturation, rates) on care organisation and system's perception by families (Likert scales)
Care givers satisfaction | Each 6 months after setting up the acquisition system in the unit
  Evaluation of carers' satisfaction with the new variables and the system's relevance in relation to their needs ("use cases" methods)
Impact on newborn's time of quiet sleep | At the end of the stay in neonatal unit, up to 10 weeks
  Quantification of the relative time of quiet sleep
Glycemia | During the stay in neonatal unit, up to 10 weeks
  Measures of physiological impact of hypo and hyperglycemias to assess the predictive value of hyperglycemia on sepsis risk
Cerebral Electrophysiology | During the stay in neonatal unit, up to 10 weeks
  Compared evaluation of data coming from Digi-NewB cohort with available data from EEG and polysomnography (impact of cerebral damages, broncho-pulmonary dysplasia)
Medium term Prognosis | During the stay in neonatal unit, up to 10 weeks
  Acquisition of magnetic resonance images (T1, T2, diffusion and cerebral perfusion arterial spin labeling) in neonatology
Prognosis evaluation | At the babies 1st and 2nd birthdays
  Assessment of the baby's neuro-development by Ages & Stages Questionnaires® (ASQ) and health related events (hospitalisation, growth...)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick PLADYS, MD, PhD, Study Director — CHU Rennes
Locations (6):
- France (6):
  - Brest University Hospital, Brest, Brittany Region
  - Angers University Hospital, Angers
  - Nantes University Hospital, Nantes
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.digi-newb.eu